CLINICAL TRIAL: NCT00805129
Title: Phase II Study of Everolimus (RAD001) in Metastatic Transitional Cell Carcinoma of the Urothelium
Brief Title: Everolimus (RAD001) in Metastatic Transitional Cell Carcinoma of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-123
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2021-12

CONDITIONS: Bladder Cancer; Metastatic Transitional Cell Carcinoma
Keywords: URETER; URINARY BLADDER; RAD001; Everolimus; Urothelium; 08-123
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Everolimus will be administered at a dose of 10 mg orally once daily continuously.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus (RAD001) is a novel oral derivative of rapamycin. Everolimus will be administered orally as a once-daily dose of 10 mg (two 5 mg tablets) continuously from study day 1 until progression of disease or unacceptable toxicity. Patients will be instructed to take Everolimus in the morning, at the same time each day. Everolimus should be taken by the patient in a fasting state or with no more than a light fat-free meal.

SUMMARY:
The purpose of this study is to learn what effects, good and/or bad, Everolimus has on advanced urothelial cancer.

The goal of this clinical research study is to learn if the study drug Everolimus can shrink or slow the growth of urothelial cancer. The safety of this drug will also be studied. The patients physical state, changes in the size of the tumor, and laboratory findings taken while on-study will help us decide if Everolimus is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis, with histological confirmation at MSKCC.
* Patients must have progressive metastatic disease. Progressive disease will be defined as new or progressive lesions on cross-sectional imaging.
* Patients must have at least one measurable site of disease (according to RECIST criteria) that has not been previously irradiated.
* Patients must have been previously treated, as defined by the following:

Treatment with at least one prior cytotoxic agent but not more than four prior cytotoxic agents. Up to four prior chemotherapy agents are allowed, since conventional chemotherapy ranges from just one drug (e.g., gemcitabine) to regimens that contain four agents (e.g., M-VAC is a four-drug regimen containing methotrexate, vinblastine, doxorubicin, and cisplatin).

* The prior therapy must have included at least one of the following: cisplatin, carboplatin, paclitaxel, docetaxel, or gemcitabine.
* The prior cytotoxic agents may have been administered in the perioperative or metastatic setting and may have been administered sequentially (e.g., first-line treatment followed by second-line treatment at time of progression) or as part of a single regimen.
* Patients must have pre-treatment tumor tissue available for analysis of m-TOR pathway markers. One paraffin block or 10 freshly-prepared unstained slides (on positively charged slides for immunohistochemistry) from the most representative single paraffin-embedded tumor tissue block. Slides from the primary tumor are preferred. If both the primary and metastatic tumor blocks are available, 10 slides from each of the sites should be submitted. If tissue from the primary tumor is not available, a paraffin block or unstained slides from a metastatic site are acceptable. Fine needle aspirates (FNAs) have insufficient tumor tissue and are not permitted.
* Age ≥ 18 years
* Karnofsky Performance Status ≥ 60%
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Adequate liver function as shown by:
* serum bilirubin ≤ 1.5 x ULN
* INR < 1.3 (or < 3 on anticoagulants)
* ALT and AST ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: If a patient's lipid values exceed either one of these criteria upon screening, the patient can only become eligible after successful initiation of appropriate lipid-lowering medication. After lipid-lowering therapy, patients must meet the same criteria - i.e. a fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN - to be eligible for study treatment
* Signed informed consent.
* Testing for hepatitis B viral load and serological markers (HBV-DNA, HBsAg, HBsAb, and HBcAb) for the following patients:

  * All patients who currently live in (or have lived in) Asia, Africa, Central and South America, Eastern Europe, Spain, Portugal, or Greece
  * Patients with any of the following risk factors:
  * Known or suspected past hepatitis B infection Blood transfusion(s) prior to 1990
* Current or prior IV drug users
* Current or prior dialysis
* Household contact with hepatitis B infected person(s)
* Current or prior high-risk sexual activity
* Body piercing or tattoos
* Mother known to have hepatitis B History suggestive of hepatitis B infection, e.g dark urine, jaundice, or right upper quadrant pain
* Additional patients at the discretion of the investigator
* Testing for hepatitis C infection (using quantitative RNA-PCR) for patients with any of the following risk factors:
* Known or suspected past hepatitis C infection (including patients with past interferon "curative" treatment)
* Blood transfusion(s) prior to 1990
* Current or prior IV drug users
* Household contact of hepatitis C infected person(s)
* Current or prior high-risk sexual activity
* Body piercing or tattoos
* Additional patients at the discretion of the investigator

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia), or patients who may require major surgery during the course of the study.
* Prior treatment with any investigational drug within the preceding 4 weeks.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent, except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg. Patients receiving these corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior to the first treatment with Everolimus. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Evidence of another active cancer, except for non-melanoma skin carcinoma, in-situ carcinoma of the cervix curatively treated, and adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is non-detectable
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Symptomatic congestive heart failure of New York Heart Association Class III or IV.
* Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease.
* Severely impaired lung function as evidenced by:

(TLC) <50% predicted, OR (FVC) <50% predicted OR, (DLCO) <40% predicted

* Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN.
* Active (acute or chronic) or uncontrolled severe infections.
* Liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis.
* A known history of HIV seropositivity.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Everolimus (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients with an active, bleeding diathesis.
* Female patients who are pregnant or breast-feeding, Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of Everolimus.
* Adults of reproductive potential who are not using effective birth control methods. Men and women of childbearing potential must be willing to use effective barrier method contraception during the trial and for at least three months thereafter. Patients are encouraged to continue barrier -method contraception for two years or longer after treatment. Hormonal contraceptives are not acceptable as a sole method of contraception
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to Everolimus (RAD001) or other rapamycins (sirolimus, temsirolimus) or to its excipients.
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-12-05 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Milowsky MI, Iyer G, Regazzi AM, Al-Ahmadie H, Gerst SR, Ostrovnaya I, Gellert LL, Kaplan R, Garcia-Grossman IR, Pendse D, Balar AV, Flaherty AM, Trout A, Solit DB, Bajorin DF. Phase II study of everolimus in metastatic urothelial cancer. BJU Int. 2013 Aug;112(4):462-70. doi: 10.1111/j.1464-410X.2012.11720.x. Epub 2013 Apr 3. PMID 23551593
- [Derived] Iyer G, Hanrahan AJ, Milowsky MI, Al-Ahmadie H, Scott SN, Janakiraman M, Pirun M, Sander C, Socci ND, Ostrovnaya I, Viale A, Heguy A, Peng L, Chan TA, Bochner B, Bajorin DF, Berger MF, Taylor BS, Solit DB. Genome sequencing identifies a basis for everolimus sensitivity. Science. 2012 Oct 12;338(6104):221. doi: 10.1126/science.1226344. Epub 2012 Aug 23. PMID 22923433
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Everolimus
Started | 46
Completed | 45
Not Completed | 1
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 46
Age, Customized [Median (Full Range); unit: years] | 66 [32 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 43
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Progression Free at 2 Months
Description: To measure the two-month PFS rate of Everolimus (RAD001) as determined by RECIST. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 45
Participants
  Progression Free | 23
  Not Progression Free | 22

2. Primary Outcome: Number of Participants Evaluated for Toxicity
Description: To determine the safety and toxicity of Everolimus (RAD001) in this patient population with toxicities being evaluated by CTCAE v3.0
Time Frame: through study completion, up to 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 46
Participants | 46

3. Secondary Outcome: Response Rate
Description: To determine the response rate of Everolimus in patients with progressive urothelial cancer who have received prior cytotoxic chemotherapy using the Response Evaluation Criteria in Solid Tumors (version 1.0). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: through study completion, up to 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 45
Participants
  Partial Response | 2
  No response | 43

4. Secondary Outcome: Proportion of Pretreatment Primary Tumor Samples With mTOR Pathway Markers
Description: To assess markers for activated mTOR pathway (including phospho-S6 and phospho-4E BP1) in all pre-treatment tissue specimens and correlate with response to treatment and PFS.
Time Frame: 25 months
Measure: Number; unit: Proportion of pretreatment primary tumor
Arm/Group | Everolimus
Number analyzed (Participants) | 45
Proportion of pretreatment primary tumor | 0.62

ADVERSE EVENTS:
Time Frame: 25 months
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 43/46
Serious Adverse Events (participants affected / at risk) | 23/46
Other Adverse Events (participants affected / at risk) | 39/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=46)
Anorexia (Metabolism and nutrition disorders) | 1
Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 2
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Edema: limb (General disorders) | 1
Enteritis (inflamm of small bowel) (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 2
Fistula, GI- Rectum (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hemorrhage, Duodenum (Gastrointestinal disorders) | 1
Hemorrhage, Urinary NOS (Renal and urinary disorders) | 1
Inf norm ANC/gr1/2 neut-Anal/perianal (Infections and infestations) | 1
Inf norm ANC/gr1/2 neut-Blood (Infections and infestations) | 1
Inf norm ANC/gr1/2 neut-Bronchitis NOS (Infections and infestations) | 1
Inf norm ANC/gr1/2 neut-Urinary(bladder) (Infections and infestations) | 1
Inf unknown ANC-Bladder(urinary) (Infections and infestations) | 1
Inf unknown ANC-Joint (Infections and infestations) | 2
Inf unknown ANC-Pneumonia(lung) (Infections and infestations) | 1
Inf unknown ANC-UTI NOS (Infections and infestations) | 2
Leukocytes (total WBC) (Investigations) | 1
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 1
Myositis (Inflamm/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 1
Pain - back (Musculoskeletal and connective tissue disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pain - Pain NOS (General disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 2
Vent arrhythmia- Ventricular tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=46)
Fatigue (General disorders) | 39
Weight loss (Investigations) | 29
Mucositis (Gastrointestinal disorders) | 24
Rash (Skin and subcutaneous tissue disorders) | 22
Constipation (Gastrointestinal disorders) | 21
Neuropathy (Nervous system disorders) | 21
Edema (General disorders) | 20
Urinary frequency (Renal and urinary disorders) | 15
Nausea (Gastrointestinal disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 10
Fever (General disorders) | 9
Diarrhea (Gastrointestinal disorders) | 7
Pain (General disorders) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Dysgeusia (Nervous system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 39
Thrombocytopenia (Investigations) | 21
Elevated Aspartate aminotransferase (Investigations) | 27
Elevated alanine aminotransferase (Investigations) | 22
Hypoalbuminemia (Metabolism and nutrition disorders) | 27
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hyperphosphatemia (Metabolism and nutrition disorders) | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hypercholesterolemia (Investigations) | 29
Hypertriglyceridemia (Metabolism and nutrition disorders) | 28
Elevated creatinine (Investigations) | 26
INR abnormal (Investigations) | 18
PTT abnormal (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT00805129/Prot_SAP_000.pdf